CLINICAL TRIAL: NCT01883765
Title: Efficacy of a Neurofeedback Treatment in Adults With ADHD: a Triple-blind Randomized Placebo-controlled Study
Brief Title: Efficacy of Neurofeedback Training in Adults With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Dr. Michael Schoenenberg, Efficacy of a Neurofeedback Treatment in Adults With ADHD: a Triple-blind Randomized Placebo-controlled Study, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCHO 1448/2-1
Record Dates: First submitted 2013-02-21; First posted 2013-06-21 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD, Neurofeedback, CBT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Color Vision Defects | interventions — Cognitive Behavioral Therapy; Psychotherapy, Group

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Neurofeedback active (Experimental): Active neurofeedback training, theta/beta-protocol
  Interventions: Behavioral: Neurofeedback active
- Neurofeedback sham (Sham Comparator): Neurofeedback training is simulated to subjects in this condition
  Interventions: Behavioral: Neurofeedback active; Behavioral: Neurofeedback sham
- Metacognitive Training (Active Comparator): Metacognitive training, cognitive behavioral therapy
  Interventions: Behavioral: Metacognitive Training

INTERVENTIONS:
Behavioral: Neurofeedback active
  Arms: Neurofeedback active; Neurofeedback sham
Behavioral: Neurofeedback sham
  Other Names: placebo neurofeedback, simulated neurofeedback
  Arms: Neurofeedback sham
Behavioral: Metacognitive Training
  Other Names: cognitive behavioral therapy, group therapy
  Arms: Metacognitive Training

SUMMARY:
Neurofeedback training (NFT) has been frequently investigated as an alternative treatment for ADHD mainly in children and adolescents. However, randomized double-blind trials that include a sham-neurofeedback control group are lacking, as well as studies examining the efficacy of NFT in adult ADHD populations. The inclusion of a sham-neurofeedback group is crucial to monitor and exclude unspecific effects.

This study aims to investigate the efficacy of NFT as compared to a sham-feedback condition and a cognitive behavioral treatment in adults with persistent ADHD.

Efficacy is assessed on several outcome parameters, such as symptom severity, neuropsychological variables (e.g., attention, memory), and EEG parameters.

ELIGIBILITY:
Inclusion criteria:

* ADHD diagnosis
* sufficient knowledge of the German language

Exclusion criteria:

* psychiatric disorder(s) lifetime (bipolar disorder, schizophrenia, schizoaffective disorder, borderline personality disorder)
* neurological disorder (e.g., epilepsy)
* current substance abuse disorder
* receives psychotherapy (e.g., CBT) or medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in ADHD symptomatology | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Conners' Adult ADHD Rating Scale (CAARS) Scores

SECONDARY OUTCOMES:
Changes in co-morbid depression scores | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Beck Depression Inventory (BDI) Scores
Changes in co-morbid anxiety scores | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  State Trait Anxiety Inventory (STAI) Scores
Changes in neuropsychological variables: Attention | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Continuous Performance Test (CPT), Errors in Omission and Errors in Commission
Changes in neuropsychological variables: Interference | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Stroop Color-Word Test, Interference scores
Changes in neuropsychological variables: Cognitive Flexibility 1 | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Test for Attentional Performance (TAP) - Flexibility, RT in ms and Errors
Changes in neuropsychological variables: Cognitive Flexibility 2 | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Inventory for Complex Attention (INKA), Items correctly performed
Changes in electrophysiological markers | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Ln-transformed theta/beta ratio
Changes in event-related potentials 1 | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Contingent Negative Variation Amplitudes
Changes in event-related potentials 2 | pre-treatment, after 8 weeks (mid-treatment), after 15 weeks (post-treatment) and after 6 months (follow-up)
  Emitted P 300 Amplitudes

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schönenberg, Dr, Principal Investigator — University Hospital Tuebingen; Martin Hautzinger, Prof. Dr., Study Chair — University Hospital Tuebingen
Locations (1):
- Universität Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schonenberg M, Wiedemann E, Schneidt A, Scheeff J, Logemann A, Keune PM, Hautzinger M. Neurofeedback, sham neurofeedback, and cognitive-behavioural group therapy in adults with attention-deficit hyperactivity disorder: a triple-blind, randomised, controlled trial. Lancet Psychiatry. 2017 Sep;4(9):673-684. doi: 10.1016/S2215-0366(17)30291-2. Epub 2017 Aug 9. PMID 28803030